CLINICAL TRIAL: NCT03525249
Title: Randomized Clinical Trial to Analyze the Efficacy of a Supplement Removed From the Internal Membrane of the Egg Shell on the Articular Pain of Diagnosed Patients of Arthrosis
Brief Title: Clinical Trial on the Articular Pain of Diagnosed Patients of Arthrosis
Acronym: FISMEH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Francisco Javier López Román, MD. PhD, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UCAM-CFE-0002
Record Dates: First submitted 2018-03-09; First posted 2018-05-15 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Comparator Membraflex 500mg (Experimental): experimental product one dose
  Interventions: Dietary Supplement: nutraceutical
- Comparator Membraflex 300mg (Experimental): experimental product two doses
  Interventions: Dietary Supplement: nutraceutical
- Placebo Comparator (Placebo Comparator): placebo product
  Interventions: Dietary Supplement: nutraceutical

INTERVENTIONS:
Dietary Supplement: nutraceutical — Subjects will consume a capsule for eight weeks

SUMMARY:
Randomized, controlled, double-blind clinical trial of three parallel branches to analyze the efficacy of a supplement extracted from the internal membrane of the egg shell on the joint pain of patients diagnosed with osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years.
* Subjects diagnosed with osteoarthritis with functional grades I-III according to the modified criteria of the American College of Rheumatology.
* Subjects must have persistent knee pain associated with osteoarthritis with an initial score of at least 30 mm in the assessment of pain according to the EVA scale.
* The subjects should not present in their treatment narcotic drugs or steroidal anti-inflammatory or immunosuppressive drugs.

Exclusion Criteria:

* Serious or terminal illnesses.
* Subjects who are currently taking glucosamine, chondroitin sulfate, collagen or hyaluronic infiltrates or any supplement indicated for joint health.
* Subjects with chronic inflammatory diseases that affect the musculoskeletal system (rheumatoid arthritis, gout, pseudo-gout, Paget's disease, chronic pain syndrome, etc.).
* Subjects with a body mass index above 32.
* Subjects with a known allergy to eggs.
* Pregnant or lactating women.
* Inability to understand informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Pain from baseline at 8 weeks | The pain will be measured by a scale twice, at the beginning and at the end of the study (after an 8 week consumption).
  analog visual scale

SECONDARY OUTCOMES:
quality of life test | it will be measured twice, once at baseline or at the end of the study after 8 weeks of use
  The quality of life of the subjects will be measured with the WOMAC test. It is a 24-item test that will measure the degree of pain on a scale of: nothing, little, enough, a lot, and a lot) when performing activities in daily life.
functional test | Twice, once at the beginning of the trial in basal conditions and once at the end after 8 weeks of consumption.
  The balance and mobility of the subjects will be measured with the Timed Up and Go Test
blood pressure | Twice, once at the beginning of the trial in basal conditions and once at the end after 8 weeks of consumption.
  the arterial pressure will be measured to the subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No